CLINICAL TRIAL: NCT06130813
Title: Effect of Increased Perioperative Communication Program on Short-Term Complications in Elective Primary Knee Arthroplasty Patients: A Randomized Controlled Trial
Brief Title: Increased Perioperative Communication Program in Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Çiğdem Canbolat Seyman, Assistant Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HU-SEYMAN-001
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Knee Arthroplasty; Postoperative Complications
Keywords: knee arthroplasty; communication program; complication; randomized controlled trial
MeSH Terms: conditions — Postoperative Complications; Communication

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Increased perioperative communication program (Experimental): The sample of the research is; it was determined as 70 patients by G. Power analysis based on the correlation coefficients in a sample study. 35 of the patients will be assigned to the intervention group (IG) and 35 to the control group (CG). Patients in the CG will receive routine perioperative care, while patients in the IG will be included in the IPCP. All patients will be followed for one month after discharge. IPCP consists of 8 informative contents such as preoperative preparations, surgical procedure, pain management, first mobilization, knee joint movements, exercise, discharge process, wound care, showering, nutrition, daily living activities, driving, sexual life, postoperative routine control, unexpected situations and etc. These informative contents will send to patients on days 7th, 4t and 1th days before the surgery and on days 1th, 2th, 3th, 5th an 7th days after surgery via whatsapp. Additionally, all participants will follow postoperative one month.
  Interventions: Other: increased perioperative communication program
- Standart of care (No Intervention): Patients in the control group will receive routine perioperative care and will follow postoperative for one month.

INTERVENTIONS:
Other: increased perioperative communication program — Thanks to this communication program, informative content (8 times) will be shared with patients.
  Arms: Increased perioperative communication program

SUMMARY:
Total knee replacement (TKA) is a surgical procedure to increase the function of the knee joint. However, in the postoperative period, it takes a long time for patients to gain independence and adapt to daily life, and they need information and support. The aim of this study is to determine the effect of the increased perioperative communication program (IPCP) in patients with TKA on early postoperative complications.

DETAILED DESCRIPTION:
Total knee replacement (TKA) is a surgical procedure to increase the function of the knee joint. However, in the postoperative period, it takes a long time for patients to gain independence and adapt to daily life, and they need information and support. The aim of this study is to determine the effect of the increased perioperative communication program (IPCP) in patients with TKA on early postoperative complications. This study was approved by the Clinical Research Ethics Committee of Ankara Bilkent City Hospital (No:E1/3573/2023). The population of this study will consist of patients who applied to Ankara Bilkent City Hospital, Orthopedics and Traumatology Outpatient Clinic due to knee osteoarthritis and who are planned to undergo elective total knee arthroplasty. Patients who are planned for elective primary unilateral knee arthroplasty, have a smartphone, are literate, have no communication problems and agree to participate in the study will be included in the study; Patients with revision total knee arthroplasty, bilateral total knee arthroplasty, speech and hearing disabilities, cognitive problems such as Alzheimer's and dementia, and patients who do not agree to participate in the study will be excluded from the study. The sample of the research is; it was determined as 70 patients by G. Power analysis based on the correlation coefficients in a sample study. 35 of the patients will be assigned to the intervention group (IG) and 35 to the control group (CG). Patients in the CG will receive routine perioperative care, while patients in the IG will be included in the IPCP. All patients will be followed for one month after discharge. IPCP consists of 8 informative contents such as preoperative preparations, surgical procedure, pain management, first mobilization, knee joint movements, exercise, discharge process, wound care, showering, nutrition, daily living activities, driving, sexual life, postoperative routine control, unexpected situations and etc. These informative contents will send to patients on days 7th, 4t and 1th days before the surgery and on days 1th, 2th, 3th, 5th an 7th days after surgery via whatsapp. Additionally, all participants will follow postoperative one month. Data will collect using Personal Information Form and Problems Experienced After Discharge Form. Data will analyze using IBM SPSS version 23.0.

ELIGIBILITY:
Inclusion Criteria:

* Elective primary unilateral knee arthroplasty planned,
* Having a smartphone,
* Literate,
* Have no communication problems and
* Agreed to participate in the study were included.

Exclusion Criteria:

* Those with revision total knee arthroplasty
* Those with bilateral total knee arthroplasty
* Those with speech and hearing disabilities and cognitive problems such as Alzheimer's and dementia
* Patients who do not agree to participate in the study will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  The investigators expect the IPCP to reduce early postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Cigdem Canbolat Seyman, PHD, Study Director — Hacettepe University
Locations (1):
- Cigdem Canbolat Seyman, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The investigators will talk about sharing data with other researchers. But it can be useful.
Supporting Information: Study Protocol, CSR
Time Frame: March 2024
Access Criteria: Data from this study can be open to all other clinical trial researchers.

REFERENCES:
- [Result] Yoon RS, Nellans KW, Geller JA, Kim AD, Jacobs MR, Macaulay W. Patient education before hip or knee arthroplasty lowers length of stay. J Arthroplasty. 2010 Jun;25(4):547-51. doi: 10.1016/j.arth.2009.03.012. Epub 2009 May 8. PMID 19427164
- [Result] Day MA, Anthony CA, Bedard NA, Glass NA, Clark CR, Callaghan JJ, Noiseux NO. Increasing Perioperative Communication With Automated Mobile Phone Messaging in Total Joint Arthroplasty. J Arthroplasty. 2018 Jan;33(1):19-24. doi: 10.1016/j.arth.2017.08.046. Epub 2017 Sep 19. PMID 29017803
- [Result] Karimi AH, Shah AK, Hecht CJ 2nd, Burkhart RJ, Acuna AJ, Kamath AF. Readability of Online Patient Education Materials for Total Joint Arthroplasty: A Systematic Review. J Arthroplasty. 2023 Jul;38(7):1392-1399. doi: 10.1016/j.arth.2023.01.032. Epub 2023 Jan 27. PMID 36716898
- [Result] Stewart MA. Effective physician-patient communication and health outcomes: a review. CMAJ. 1995 May 1;152(9):1423-33. PMID 7728691
- [Result] Clarke HD, Timm VL, Goldberg BR, Hattrup SJ. Preoperative patient education reduces in-hospital falls after total knee arthroplasty. Clin Orthop Relat Res. 2012 Jan;470(1):244-9. doi: 10.1007/s11999-011-1951-6. PMID 21691907